CLINICAL TRIAL: NCT00558051
Title: Phase I Evaluation of Semi-continuous Alpha-type-1 Dendritic Cell-based Vaccines in Patients With Metastatic Colorectal Cancer
Brief Title: Alpha-type-1 Dendritic Cell-based Vaccines in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pawel Kalinski (Other)
Responsible Party: Sponsor-Investigator, Pawel Kalinski, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 05-063
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intradermal administration (Active Comparator): Intradermal administration
  Interventions: Biological: DC-based vaccine
- Intranodal administration (Active Comparator): Intranodal administration
  Interventions: Biological: DC-based vaccine
- Intralymphatic infusion (Active Comparator): Intralymphatic infusion
  Interventions: Biological: DC-based vaccine

INTERVENTIONS:
Biological: DC-based vaccine — Each patient will receive four courses of vaccination with 2 million tumor-loaded DCs at week 0, 4, 8, and 12. A course consists of 4 intradermal injections once a day for 4 days.
  Arms: Intradermal administration
Biological: DC-based vaccine — Each patient will receive four courses of vaccination with 2 million tumor-loaded DCs at week 0, 4, 8, and 12. A course consists of 1 intranodal injection.
  Arms: Intranodal administration
Biological: DC-based vaccine — Each patient will receive four courses of vaccination with 2 million tumor-loaded DCs at week 0, 4, 8, and 12. A course consists of a 4-day intralymphatic infusion.
  Arms: Intralymphatic infusion

SUMMARY:
The purpose of this study is to evaluate the administration, safety and immunologic effectiveness of an experimental vaccine for colorectal cancer patients.

DETAILED DESCRIPTION:
Dendritic cell (DC)-based vaccination, usually administered by a traditional intradermal route, is a new treatment option for cancer patients. While the previous DC-based vaccination trials have shown the safety of this approach and its ability to induce objective clinical responses, the overall efficacy of DC-based vaccines is still disappointing (Rosenberg et al., 2004). We hypothesize that the two likely causes of such limited clinical activity are: A) suboptimal type of DCs used as a vaccine and B) suboptimal modes of use of such vaccines that do not allow the vaccinated patients to fully benefit from DC biology.

We will conduct a pilot evaluation of the therapeutic vaccination with DC1s loaded with autologous tumor material, in patients with metastatic colorectal cancer that have been resected to no or minimal evidence of disease.The proposed evaluation of the novel intralymphatic route of DC-based vaccination will allow us to administer the vaccine in a way that is more physiologic with respect to the kinetics of antigen appearance to the lymph nodes and is feasible to be performed in repetitive fashion, without damaging local lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic colorectal cancer with minimal evidence of disease or resectable metastases (to include extra-hepatic metastases).
* Availability of metastatic tumor material, from hepatic metastasis and additional sites, that can be resected under sterile conditions for autologous vaccine preparation (not all tumors harvested will be of sufficient quantity or quality to make vaccine, therefore some subjects may not receive vaccine).
* No chemotherapy, radiotherapy, major surgery, or biologic therapy for their malignancy in the 4 weeks prior to the vaccine administration and must have recovered from all side effects.
* An ECOG performance standard of 0, 1 or 2.
* Adequate hepatic function as evidenced by bilirubin < 2.0 mg/dL and a PT < 2 seconds of the upper limit of normal.
* Age equal to 18 years or older and greater than 30 kg.
* Platelet counts greater than 100,000, a hematocrit > 27.0, a white blood count > 3000/µl, and a creatinine less than or equal to 1.5 mg/dL or a creatinine clearance of > 60 mL/min.
* Aware of the neoplastic nature of his/her illness, the experimental nature of the therapy, alternative treatments, potential benefits and risks, and willing to sign an informed consent.
* Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

* Subjects currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 4 weeks after removal from immunosuppressive treatment. Subjects on maintenance steroids because of adrenal insufficiency are eligible.
* Subjects with severely abnormal liver function tests [AST (SGOT), ALT (SGPT), GGT, Alk.Phos, LDH, and total bilirubin greater than 2 X ULN]
* Subjects with uncontrolled pain.
* Subjects with active autoimmune disease, positive serology for HIV, HBV, or HCV (testing will be performed with FDA licensed blood donor tests).
* Subjects with concurrent additional malignancy (with exception of non-melanoma skin cancers and carcinoma in situ of the cervix).
* Subjects who are allergic to or develop an allergy to heparin.
* Subjects who are pregnant.
* Subjects who have sensitivity to drugs that provide local anesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is to evaluate the feasibility and safety of semi-continuous intralymphatic vaccination dendritic cells. | 4 to 14 weeks

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the immunity results from either single injections or semi-continuous infusion, intradermal or intranodal, administered immunization with the DC vaccine for colorectal cancer (CRC) patients. | 4 to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David L. Bartlett, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Radomski M, Zeh HJ, Edington HD, Pingpank JF, Butterfield LH, Whiteside TL, Wieckowski E, Bartlett DL, Kalinski P. Prolonged intralymphatic delivery of dendritic cells through implantable lymphatic ports in patients with advanced cancer. J Immunother Cancer. 2016 Apr 19;4:24. doi: 10.1186/s40425-016-0128-y. eCollection 2016. PMID 27096100